CLINICAL TRIAL: NCT01652781
Title: A Randomized, Phase II, Comparative Study With a Parallel Control for Evaluating the Efficacy and Safety of 5-day Azacitidine for Patients With Lower-risk Myelodysplastic Syndrome
Brief Title: 5 Day Versus 7 Day Azacitidine in Lower Risk Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Yoo-Jin Kim, Associate Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VZ-MDS-PI-0267
Record Dates: First submitted 2012-07-11; First posted 2012-07-30 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: myelodysplastic syndrome; azacitidine; dosing schedule
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-day arm (Experimental): azacitidine 75mg/m2 subcutaneously for 7 days every 28 days + best supportive care
  Interventions: Drug: Azacitidine
- 7-day arm (Active Comparator): azacitidine 75mg/m2 subcutaneously for 5 days every 28 days + best supportive care
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — 5-day arm: azacitidine 75mg/m2 subcutaneously for 7 days every 28 days + best supportive care 7-day arm: azacitidine 75mg/m2 subcutaneously for 5 days every 28 days + best supportive care
  Other Names: vidaza

SUMMARY:
Approved dosing schedule of azacitidine for myelodysplastic syndrome (MDS) is 75 mg/m^2/day subcutaneous for 7 consecutive days every 28 days, which is based on the data from standard chemotherapy regimen and a Phase I safety clinical trial. Since the optimal dosage of this drug has not been found yet, it remains as a subject of clinical study that needs to be examined. If initial toxicity is minimized by developing dosage/regimen that replaces the standard therapy, it will be possible to provide continuous treatment with increased convenience by patients and treating physicians as well as improvement for safety in elderly patients or those with serious cytopenia. In addition, it is expected to lead to a better response by strictly keeping a treatment schedule.

Recent US study showed that 5-day regimen showed similar treatment results, but retrospective data from Spain showed lower response rate in 5-day regimen. Considering the recent circumstances around dosage and schedule of azacitidine in lower risk MDS, a Phase II clinical trial is planned in lower risk MDS patients in order to explore the efficacy in 5-day treatment by comparing prospectively with 7-day standard regimen.

DETAILED DESCRIPTION:
* Using block randomization, subjects of Low or intermediate (INT)-1 patients will be equally allocated to the following two types of regimens.

  1. Group A: azacitidine 75mg/m^2 subcutaneously for 7 days every 28 days + best supportive care
  2. Group B: azacitidine 75mg/m^2 subcutaneously for 5 days every 28 days + best supportive care
* The study drug, azacitidine, is provided free of charge by Celgene until disease progression or relapse after response, or intolerable toxicity occurs in clinical study subject, or informed consent is withdrawn.
* No crossover between arms is allowed.
* Dose escalation in this study is not allowed; on the contrary, dose reduction or dose delay is possible based on adverse events and hematologic recovery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria in order to be enrolled in this clinical trial: Patients who have been diagnosed with MDS by the FAB criteria and belong to Low or INT-1 risk by the IPSS classification will be enrolled in this study. For the purpose of analysis, chronic myelomonocytic leukemia (CMML) patients with less than 5% of myeloblasts are also classified by the IPSS risk classification. Secondary or treatment-related MDS is allowed, but recurrent or persistent MDS after stem cell is not applicable. The enrolled patients should have anemia (hemoglobin < 10.0g/dL), transfusion dependence, thrombocytopenia (less than 100×10^9/L), or absolute neutrophil count less than 1.80×10^9/L.
* 18 years of age or older
* Life expectancy of at least 12 months
* ECOG performance status 2 or less
* Serum creatinine less than 1.5 times the upper limit of normal (ULN) level of the investigating institution
* Serum bilirubin less than 2.0 times the upper limit of normal (ULN) level of the investigating institution
* AST, ALT, and alkaline phosphatase less than 3 times the upper limit of normal (ULN) level of the investigation institution
* Patients who can have informed consent and signed the informed consent form
* Male patients who have a female partner of childbearing potential must agree to use two types of effective contraceptive methods during the study and for 30 days following the last dose.
* Females of childbearing potential (FCBP) must satisfy the following criteria: must agree to use the contraceptive method (oral contraceptives, injectables, hormonal implants; tubal ligation; intra uterine device; spermicidal contraceptives, the sterilized partner) approved by the physician during azacitidine treatment and for 3 months following the last dose, and must have a negative result of serum pregnancy test that was performed within 72 hours prior to starting study drug therapy.

Exclusion Criteria:

* Any coexisting major illness or organ failure
* HIV positive, or active hepatitis B or C infection
* Uncontrolled acute infection
* Uncontrolled hemorrhage
* Pregnant or lactating
* Known or suspected hypersensitivity to azacitidine
* Patients diagnosed with malignant hepatic carcinoma or malignant disease within the past 12 months (except in situ carcinoma without complication, cervical or breast intraepithelial neoplasia, or other local malignant carcinoma that is likely to be treated by surgical removal or radiotherapy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate by modified IWG 2006 response criteria | After 6 cycles of treatment up to 25-49 weeks
  Overall response rate is evaluated by assessing the percentage of patients with response (complete remission (CR), partial remission (PR), bone marrow CR, and hematologic improvement), response period, and transfusion requirement. Best response during at least 6 cycles of treatment will be assessed if there is no treatment failure or disease progression within 6 cycles of treatment. For patients who can keep the 4 week interval the Time Frame will be 25 weeks. The cycle interval can be extended up to 8 weeks which makes 49 weeks the maximum Time Frame.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | After each course of treatment up to 25-49 weeks
  •Safety and tolerability profile of 5-day azacitidine in comparison with 7-day regimen. For patients who can keep the 4 week interval the Time Frame will be 25 weeks. The cycle interval can be extended up to 8 weeks which makes 49 weeks the maximum Time Frame.
Cytogenetic response rate by IWG 2006 response criteria | After 6 cycles of treatment up to 25-49 weeks
  •Cytogenetic response of of 5-day azacitidine in comparison with 7-day regimen. For patients who can keep the 4 week interval the Time Frame will be 25 weeks. The cycle interval can be extended up to 8 weeks which makes 49 weeks the maximum Time Frame.

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Jin Kim, MD, PhD, Principal Investigator — Division of hematology, Department of Internal Medicine, Catholic Blood and Marrow Transplantation Center, Seoul St. Mary's Hospital
Locations (3):
- South Korea (3):
  - Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul